CLINICAL TRIAL: NCT00178893
Title: CellzDirect: Hepatocellular Research Registry
Brief Title: Hepatocellular Research Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sunil Geevarghese, MD, MSCI, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 040220
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Hepatocytes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hepatocytes
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry of human hepatocytes (liver cells) for research purposes.

DETAILED DESCRIPTION:
Patients scheduled for partial hepatectomy/liver surgery are asked permission to use their discarded liver tissue for purposes of studying:

1. how drugs/medicines affect the liver and
2. the effects of storing liver cells in the cold or freezing.

ELIGIBILITY:
Inclusion Criteria:

* Persons undergoing partial hepatectomy/liver surgery for any reason.

Exclusion Criteria:

* Persons with known HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* A diagnosis of hepatocellular carcinoma without negative serologies
* A diagnosis of cholangiocarcinoma, where the total bilirubin has ever been greater or equal to 3.0
* The presence of a biliary drainage tube
* Active sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient having liver resection operation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K Geevarghese, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States